CLINICAL TRIAL: NCT07251621
Title: Evaluation of the Application Effect of a Surgical Navigation System in HoLEP Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Qing Yuan, Professor, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S202403101
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Benign Prostate Hypertrophy(BPH)
Keywords: Benign Prostate Hypertrophy; holmium laser enucleation of the prostate; Surgical Navigation System
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- use of the 3D imaging-assisted surgical navigation system during surgery (Experimental): Based on the use of the 3D imaging-assisted surgical navigation system during surgery, patients were divided into an Observation group and a Control group
  Interventions: Procedure: use the 3D imaging-assisted surgical navigation system during surgery

INTERVENTIONS:
Procedure: use the 3D imaging-assisted surgical navigation system during surgery — Based on the use of the 3D imaging-assisted surgical navigation system during surgery, patients were divided into an Observation group and a Control group.

SUMMARY:
3D imaging-assisted surgical navigation system was established using the following specific procedures: 1) Prostate MRI Acquisition and 3D Reconstruction: patient prostate MRI images are acquired, and professional engineers complete 3D reconstruction; 2) Data Import to Diagnostic Ultrasound System: Reconstructed prostate MRI images and P-3DRI (Prostate 3D Reconstruction Image) data are imported into the Diagnostic Ultrasound system; 3) Transrectal Ultrasound Probe Placement: The transrectal ultrasound probe is secured to a dedicated holder. The probe is inserted into the patient's rectum to locate the prostate. After manual adjustment to optimize imaging, the holder is fixed in position; 4) Initial Position Registration: The Diagnostic Ultrasound system integrates prostate MRI, P-3DRI, and real-time ultrasound images. Spatial correspondence between P-3DRI and the actual prostate position is established using real-time ultrasound; 5) Cystoscope-Electromagnetic Navigation Assembly: A self-designed electromagnetic navigation connector links the electromagnetic sensor to the cystoscope. The ultrasound probe is simultaneously equipped with an electromagnetic sensor; 6) Real-time Spatial Tracking and Fusion: The electromagnetic navigation module tracks spatial positions of surgical instruments and the ultrasound probe. These positions are fused with real-time ultrasound coordinates.

Through the above steps, the relative position between surgical instruments and the prostate is displayed in real time, achieving intraoperative navigation. All procedures were performed by the same Associate Chief Physician at our medical center. Based on the use of the 3D imaging-assisted surgical navigation system during surgery, patients were divided into an Observation group and a Control group.

ELIGIBILITY:
Inclusion Criteria:

* 1) Clinically diagnosed BPH patients with LUTS; 2) Voluntarily participated in the clinical trial and provided written informed consent; 3) Met the surgical intervention indications outlined in the 2019 'Chinese Guidelines for Diagnosis and Treatment of Urological Diseases'; 4) Completed preoperative BPH evaluations, including International Prostate Symptom Score (IPSS) and Quality of Life (QoL) assessment.

Exclusion Criteria:

* 1) Refusal to participate in the clinical trial; 2) Presence of severe uncontrolled medical conditions or psychiatric disorders; 3) Cognitive impairment impeding normal communication.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
postoperative complications | month 1；month 3；
  Urinary Incontinence (Defined as an International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) score ≥ 1), Urethral Stricture (Defined as recurrence of dysuria or narrowed urine stream postoperatively, confirmed by cystoscopy)

CONTACTS AND LOCATIONS:
Locations (1):
- ChinaPLAGH, Beijing, Haidian, China

IPD SHARING:
Plan to Share IPD: No